CLINICAL TRIAL: NCT02950610
Title: Breath Analysis Using an Electronic Nose in Non Alcoholic Fatty Liver Disease (BEN) Study
Brief Title: Breath Analysis Using an Electronic Nose in Non Alcoholic Fatty Liver Disease
Acronym: BEN
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: University of Strathclyde (Other); University of Amsterdam (Other)
Responsible Party: Sponsor
Other Study IDs: 165914
Record Dates: First submitted 2016-01-13; First posted 2016-11-01 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2016-10

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Electronic nose; Non invasive diagnosis of NAFLD; NAFLD; exhaled breath analysis; Volatile organic compounds
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool, urine and blood sample for predetermined Non-DNA analysis. Intestinal microbial identification with 16s RNA sequencing
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy: Healthy volunteer: self-declared healthy individual (no known illness or medications) with Normal BMI
  Interventions: Device: Breath analysis - electronic signature "Breath-print"
- Nonalcoholic steatohepatitis: NAFLD without cirrhosis: Metabolic syndrome with known liver disease (NAFLD, excluding other coexisting liver condition) without cirrhosis
  Interventions: Device: Breath analysis - electronic signature "Breath-print"
- NAFLD Cirrhosis: NAFLD cirrhosis: well characterised NAFLD compensated cirrhosis (Child's A-B)
  Interventions: Device: Breath analysis - electronic signature "Breath-print"

INTERVENTIONS:
Device: Breath analysis - electronic signature "Breath-print" — Patients and Healthy volunteers ( as defined in 3 cohorts) will breath into disposable, once-use only bacterial filter channeled into electronic device comprising on sensors capable to reacting to organic compounds. Breathing manoeuvre will be simple, non-exertional and relaxed. 2 breathing manoeuvres will be performed and sensor responses will be captured.

SUMMARY:
The purpose of this is to analyse human exhaled breath by means of a device called electronic nose(eNose) in patients with non-alcoholic fatty liver disease (NAFLD) as a way to non-invasive assessment of liver disease.This device is medically adapted and clinically validated in patients with lung conditions.

DETAILED DESCRIPTION:
Human exhaled breath contains over 3000 volatile organic compounds (VOCs) that vary in relative concentration in health and disease. Metabolic disorders affecting the liver, such as NAFLD, produce disproportionate organic compounds produced as a by-product of metabolism and thus expired in exhaled breath, excreted in urine and detectable in blood. NAFLD prevalence is increasing and has reached epidemic proportions affecting 90% of obese adults and 22%-53% of obese children.Liver biopsy is the gold standard in diagnosing NAFLD, but it is unpleasant and can lead to complications. There is an unmet need to develop a non-invasive method of assessing liver disease. Comon Invent (Delft, Netherlands) together with the respiratory department at the Amsterdam Medical Centre (AMC), University of Amsterdam, have adapted the electronic nose known as SpiroNose as a prototype device for clinical use. Sensitive electronic sensors detect molecules in breath and generate signals. Complex algorithms and analytical technics allow pattern recognition of breath samples from different subjects. Well charaterised patients will be selected into clinical categories of non-alcoholic fatty liver disease with and without cirrhosis and be compared with healthy individuals.

Edinburgh will be the only site conducting this study. In addition to exhaled breath analysis, blood and urine will be collected to study the end products of metabolism.Furthermore, stool and urine collected from some subjects will be analysed to understand the role of gut bacteria in fermentation, metabolic products as a result cause VOC production.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals with no known or self declared medical illness with BMI (body mass index) within normal range (18.5-25)
* Non alcoholic fatty liver disease without cirrhosis
* Compensated (no evidence of ascites, encephalopathy) NAFLD cirrhosis; assessed by scoring system - Child's Pugh

Exclusion Criteria:

* Ongoing or recent (within last 6months) alcohol consumption more than 21 units per week for males and 14 units per week for females.
* BMI > 40
* Chronic respiratory disease e.g. Chronic obstructive pulmonary disease (COPD), asthma, interstitial fibrosis
* Use of antibiotics within last 4 weeks of sample collection and inflammatory bowel disease, irritable bowel syndrome, celiac sprue, or other chronic inflammatory diseases of the intestines (for intestinal microbiome analysis)
* Other known liver disease e.g. Primary Biliary Cholangitis/cirrhosis (PBC), Alcoholic liver disease (ALD), Autoimmune and hepatitis
* Inability to provide informed consent.
* Participation in other clinical intervention/drug trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All eligible patients will have to consent to the study. The study population will consist of participants aged between 18 and 75 years old in the following cohorts (Healthy individuals, Non-alcoholic steatohepatitis (non-cirrhotic) and compensated Non-alcoholic liver cirrhosis). Each cohort will have 30 patients. There will be an equal number of participants for the healthy control group. In summary, the investigators aim to recruit 30 subject in the patient cohorts and 30 in healthy, totaling a number of 90 in the study
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Characterise the electronic signature "breath-print" in pre-defined cohorts | 12 months
  Identify disease specific electronic nose wave pattern
Characterisation of exhaled breath composition | 12 months
  Molecular characterisation of breath volatile organic compounds through Gas Chromatography and Mass Spectrometry

SECONDARY OUTCOMES:
Profiling intestinal microbiome and assessing end-metabolic products in urine | 12 months
  Demonstrate dysbiosis in stool microbial and characterise metabolic products in urine of cohorts studied

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Hayes, MD,PhD,FRCPE, Principal Investigator — Centre for liver and digestive disorder, Royal Infirmary of Edinburgh, Edinburgh, EH16 4SA
Locations (1):
- Clinical Research Facility - Wellcome Trust, Royal Infirmary Site, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not shared. Participants will be identified as a part of pre-defined cohort as categorised clinically.

REFERENCES:
- [Result] Wlodzimirow KA, Abu-Hanna A, Schultz MJ, Maas MA, Bos LD, Sterk PJ, Knobel HH, Soers RJ, Chamuleau RA. Exhaled breath analysis with electronic nose technology for detection of acute liver failure in rats. Biosens Bioelectron. 2014 Mar 15;53:129-34. doi: 10.1016/j.bios.2013.09.047. Epub 2013 Sep 30. PMID 24135544
- [Result] de Vries R, Brinkman P, van der Schee MP, Fens N, Dijkers E, Bootsma SK, de Jongh FH, Sterk PJ. Integration of electronic nose technology with spirometry: validation of a new approach for exhaled breath analysis. J Breath Res. 2015 Oct 15;9(4):046001. doi: 10.1088/1752-7155/9/4/046001. PMID 26469298
- [Result] Probert CS, Ahmed I, Khalid T, Johnson E, Smith S, Ratcliffe N. Volatile organic compounds as diagnostic biomarkers in gastrointestinal and liver diseases. J Gastrointestin Liver Dis. 2009 Sep;18(3):337-43. PMID 19795029
- [Result] Wu GD, Lewis JD, Hoffmann C, Chen YY, Knight R, Bittinger K, Hwang J, Chen J, Berkowsky R, Nessel L, Li H, Bushman FD. Sampling and pyrosequencing methods for characterizing bacterial communities in the human gut using 16S sequence tags. BMC Microbiol. 2010 Jul 30;10:206. doi: 10.1186/1471-2180-10-206. PMID 20673359
- [Derived] Sinha R, Gillespie SL, Brinkman P, Bassett P, Lockman KA, Jaap AJ, Fallowfield JA, Hayes PC, Plevris JN. Volatomics for Diagnosis and Risk Stratification of MASLD: A Proof-Of-Concept Study. Aliment Pharmacol Ther. 2025 Jul;62(2):180-192. doi: 10.1111/apt.70176. Epub 2025 May 20. PMID 40391721
- [Derived] Sinha R, Lockman KA, Homer NZM, Bower E, Brinkman P, Knobel HH, Fallowfield JA, Jaap AJ, Hayes PC, Plevris JN. Volatomic analysis identifies compounds that can stratify non-alcoholic fatty liver disease. JHEP Rep. 2020 Jun 15;2(5):100137. doi: 10.1016/j.jhepr.2020.100137. eCollection 2020 Oct. PMID 32775974